CLINICAL TRIAL: NCT06876064
Title: National Cohort of Subjects at Risk of Developing Rheumatoid Arthritis
Acronym: PROMESS_1
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Nantes University Hospital (Other); Assistance Publique Hopitaux De Marseille (Other); UNIVERSITY HOSPITAL, ORLEANS (Unknown); Bicetre Hospital (Other); Saint Antoine University Hospital (Other); Groupe Hospitalier Pitie-Salpetriere (Other); University Hospital, Brest (Other); Assistance Publique - Hôpitaux de Paris (Other); University Hospital, Bordeaux (Other); Hôpital Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL24_0015; Eudra CT/ID-RCB (Other: 2024-A01176-41)
Record Dates: First submitted 2024-12-24; First posted 2025-03-14 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: at-risk; ACPA; Rheumatoid arthritis; Exposome; Prediction
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Hematologic Tests; Urinalysis; Wettability; Radiography, Panoramic; Referral and Consultation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection:
  A total of 60 ml of blood will be collected while fasting, using the following tubes: one PAXGene Blood RNA Tube, one PAXGene Blood DNA Tube, five 5 mL serum tubes, five 5 mL EDTA tubes and one 2 mL EDTA tube for microbiota DNA analysis.
  Urine collection:
  Urine will be collected, while fasting and after the administration of lactulose/ mannitol to assess intestinal permeability.
  Stool collection:
  Stool samples will be collected either at the hospital or at home using a dedicated kit.
  Saliva collection:
  5 ml of saliva will be collected and saliva microbiome DNA will be collected using an OMNIgene Oral kit.
  Induced expectoration:
  Induced sputum is collected after the inhalation of salbutamol (hypertonic aerosol).
  Hair sampling:
  Hair samples will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: A total of 50 subjects will be recruited: individuals with ACPA≥2 N and clinically suspect arthralgia (CSA criteria ≥4) or those with ACPA≥N and rheumatoid factor≥2N along with clinically suspect arthralgia (CSA criteria ≥4). These subjects have an estimated 50% risk of progression to RA within 2 years.
  Interventions: Biological: Blood test; Biological: Urine test; Other: stool collection; Other: saliva collection; Other: Induced expectoration; Other: Hair and nails sampling; Other: Schirmer test; Radiation: Ultrasound of hands and feet; Radiation: MRI Contrast; Other: Patient questions; Diagnostic Test: Dental panoramic X-ray; Other: Consultation with a psychologist in certain centers; Other: Measurement of heart rate variability.
- Group 2: A total of 50 subjects will be recruited: individuals with ACPA≥2 N who do not meet the criteria for clinically suspect arthralgia (CSA criteria <4) or those with ACPA≥N and rheumatoid factor≥2N who also do not meet the criteria for clinically suspect arthralgia (CSA criteria <4). These subjects have an estimated 30% risk of progression to RA within 2 years.
  Interventions: Biological: Blood test; Biological: Urine test; Other: stool collection; Other: saliva collection; Other: Induced expectoration; Other: Hair and nails sampling; Other: Schirmer test; Radiation: Ultrasound of hands and feet; Radiation: MRI Contrast; Other: Patient questions; Diagnostic Test: Dental panoramic X-ray; Other: Consultation with a psychologist in certain centers; Other: Measurement of heart rate variability.
- Group 3: A total 25 subjects will be recruited: asymptomatic subjects (CSA criteria <4) with a family history of RA in a first-degree relative (negative controls).
  Interventions: Biological: Blood test; Biological: Urine test; Other: stool collection; Other: saliva collection; Other: Induced expectoration; Other: Hair and nails sampling; Other: Schirmer test; Radiation: Ultrasound of hands and feet; Radiation: MRI Contrast; Other: Patient questions; Other: Consultation with a psychologist in certain centers; Other: Measurement of heart rate variability.
- Group 4: A total of 25 subjects will be recruited: individuals with RA diagnosed at polyarthritis onset (diagnosis <6 months) who have not yet been treated, with ACPA≥2 N or ACPA≥N and rheumatoid factor≥2N (positive controls).
  Interventions: Biological: Blood test; Biological: Urine test; Other: stool collection; Other: saliva collection; Other: Induced expectoration; Other: Hair and nails sampling; Other: Schirmer test; Radiation: Ultrasound of hands and feet; Radiation: MRI Contrast; Other: Patient questions; Diagnostic Test: Dental panoramic X-ray; Other: Consultation with a psychologist in certain centers; Other: Measurement of heart rate variability.

INTERVENTIONS:
Biological: Blood test — A total of 60 ml of blood will be collected while fasting, using the following tubes: one PAXGene Blood RNA Tube, one PAXGene Blood DNA Tube, five 5 mL serum tubes, five 5 mL EDTA tubes and one 2 mL EDTA tube for microbiota DNA analysis.
Biological: Urine test — Urine will be collected, while fasting and after the administration of lactulose/ mannitol to assess intestinal permeability.
Other: stool collection — Stool samples will be collected either at the hospital or at home using a dedicated kit.
Other: saliva collection — 5 ml of saliva will be collected and saliva microbiome DNA will be collected using an OMNIgene Oral kit.
Other: Induced expectoration — inhalation of salbutamol, measurement of peak expiratory flow by screening spirometry (15 min later), inhalation of a hypertonic aerosol for 3 periods of 7 min. At the end of each inhalation period, the induced sputum is collected and the peak expiratory flow is measured to prevent possible bronchospasms
Other: Hair and nails sampling — Hair and nails samples will be collected.
Other: Schirmer test — To assess of tear secretion
Radiation: Ultrasound of hands and feet — To assess the risk of RA in high-risk subjects by evaluating for synovitis, tenosynovitis, or intermetatarsal-phalangeal bursitis.
Radiation: MRI Contrast — MRI of the dominant or painful hand will be performed to assess the risk of RA in high-risk subjects.
Other: Patient questions — Self-questionnaires will assess factors such as ethnic origin, family history of RA, diet, physical activity, exposure to toxic substances, pollution, occupational exposures, psychological and clinical factors.
Diagnostic Test: Dental panoramic X-ray — Performed as part of routine care to assess dental health
  Groups: Group 1; Group 2; Group 4
Other: Consultation with a psychologist in certain centers — The short-CTQ will be completed during this consultation, only in centers offering consultations with a psychologist.
Other: Measurement of heart rate variability. — The patient will wear a belt throughout the visit 1. At the end of the day, the heart rate variability data measured by the belt will be recorded in the CRF (RR interval, heart rate variability SDNN, RMSSD, and LF/HF sympathovagal balance).

SUMMARY:
PROMESS 1 is a multicenter cohort interventional study aiming at analyzing the factors associated with the risk of developing clinical arthritis among exposures or combinations of exposures in patients at risk of rheumatoid arthritis (RA), as they have high levels of anti-citrullinated peptides autoantibodies (ACPA ≥2 N).

The primary endpoint is the occurrence of clinical arthritis confirmed by ultrasound at two years of following for the subject's groups at risk of RA.

This may be explained by the following exposures or combinations of exposures: smoking, occupational exposure, physical activity, diet, hormonal exposure, drug exposure, trauma and psychological stress.

Other factors may also explain the occurrence of clinical arthritis:

* Other symptoms
* Comorbidities, medical history, drug exposures
* Current biology: ACPA levels, rheumatoid factor levels and isotypes, CRP levels at baseline, etc.
* Ultrasound and MRI abnormalities.

DETAILED DESCRIPTION:
This is a multicenter interventional cohort study. The goal of this cohort is to analyze the factors associated with the risk of developing clinical arthritis, considering individual or combined exposures, in patients at high risk of rheumatoid arthritis (RA).

Four groups of adults will be included:

* Group 1: 50 subjects at very high risk of RA: ACPA≥2 N or (ACPA>N and rheumatoid factor≥2 N) + presence of clinically suspicious arthralgia (CSA criteria ≥4)
* Group 2: 50 subjects at high risk of RA: ACPA≥2 N or (ACPA>N and rheumatoid factor≥2 N) without clinically suspicious arthralgia (CSA criteria <4)
* Group 3: 25 asymptomatic subjects, 1st degree relatives of subjects with RA (negative controls)
* Group 4: 25 patients with early RA prior to any disease-modifying therapy (positive controls) Patients in the control groups will be included based on the same age and sex as patients in the risk groups (1 & 2) in the recruiting center.

The primary endpoint is the occurrence of clinical arthritis, confirmed by ultrasound, after two years of follow-up in the at-risk RA groups (Groups 1 & 2).

This may be explained by the following exposures or their combinations: smoking, occupational exposure, physical activity, diet, hormonal exposure, drug exposure, trauma and psychological stress...

Other factors that may contribute to the occurrence of clinical arthritis include:

* Clinical elements and questionnaires assessing the other symptoms of the individuals (PRO) (subjective clinical suspicion of arthralgia CSA, painful joints at inclusion, BMI, stool consistency, functional respiratory signs, etc.)
* Comorbidities and antecedents via CNAM pathology mapping and drug exposure via data on dispensing in towns from the SNDS
* Current biology: ACPA levels, rheumatoid factor levels and isotypes, CRP levels at baseline, etc.
* Ultrasound and MRI abnormalities.

The controls groups (groups 3&4) will allow for a cross-sectional analysis, comparing at-risk RA subjects with healthy individuals who share the same genetic background. They will have a single visit at baseline without follow-up.

However, the at-risk RA groups (groups 1 & 2) will have four visits (M0, M6, M12 et M24). In addition to routine care examinations performed in RA risk situations, subjects will undergo blood and stool sample collection at baseline and at one year.

All subjects regardless of group, will undergo the following baseline assessments: MRI of the dominant hand or painful hand, a lactulose absorption test (to assess intestinal permeability), hair and saliva collection, a Schirmer test, and, in some centers, an induced sputum test (to assess pulmonary mucosa). Ultrasound of the hands and feet, as well as specific questionnaires assessing the exposome, will be conducted at all visits.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years old
* Group 1: Individuals with high risk of RA (ACPA ≥ 2N or ACPA ≥ N and rheumatoid factor ≥ 2N) and clinical signs of arthralgia (CSA criteria ≥ 4).
* Group 2: High-risk individuals (ACPA ≥ 2N or ACPA ≥ N and rheumatoid factor ≥ 2N) without clinical arthralgia (CSA criteria < 4).
* Group 3: First-degree relatives of RA patients (no symptoms, negative controls).
* Group 4: Newly diagnosed untreated RA patients (ACPA ≥ 2N or ACPA ≥ N and rheumatoid factor ≥ 2N) (positive controls).

Exclusion Criteria:

* Groupe1-2-3:

  • Presence of clinical joint swelling (synovitis) at the time of inclusion and previously noted by a doctor
* All groups:

  * Taking current or past background treatment for RA, even for another indication
  * Corticosteroid therapy ≥10 mg at baseline and in the previous week
  * Presence of another connective tissue disease (Sjögren's, dermatomyositis, scleroderma, Sharp syndrome, etc.)
  * Subject unable to read and/or write
  * Inability to follow the patient during the study period
  * Failure to obtain consent
  * Non-affiliation to a social security scheme,
  * Persons placed under legal protection, under curatorship or under guardianship
  * Pregnant or breastfeeding women
  * Person participating in another intervention research including an
  * exclusion period still in progress

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients will be recruted during consultation or hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Risk of developing clinical arthritis | From the baseline to the end of the follow-up at 2 years
  To analyze the factors associated with the risk of developing clinical arthritis confirmed by ultrasound among exposures or combinations of exposures in patients at high risk of RA.

SECONDARY OUTCOMES:
Quantitative difference in Food Frequency Questionnaire (FFQ) between the 4 groups of subjects included, varying from never or rarely to daily or multiple times per day. | At baseline
Quantitative difference in National Observatory for Physical Activity and Sedentariness -Physical Activity Questionnaire (ONAPS-PAQ) expressed in MET (Metabolic Equivalent of Task) per week between the 4 groups of subjects included. | At baseline
Quantitative difference in patient-reported exposure outcome Alcohol and Substance Involvement Screening Test (ASSIST) score between the 4 groups of subjects included. | At baseline
  The score varies from 0 to 36 to each substance with higher score indicates greater substance-related risk and the need for stronger intervention strategies.
Quantitative difference in Fagerström Test for Nicotine Dependence (FTND) score between the 4 groups of subjects included. | At baseline
  The score varies from 1 to 6 with higher score indicate greater nicotine dependence.
Compare the exposure to pollution between the 4 groups of subjects included. "Exposure to pollution will be assessed by cross-referencing residential addresses with the Chimère database. | At baseline
Qualitative difference in a self-report integrated questionnaire for diagnosis of all functional gastrointestinal disorders in adults between the 4 groups of subjects included. | At baseline
Quantitative difference in patient-reported Francis score for Irritable Bowel Syndrome (IBS) between the 4 groups of subjects included. | At baseline
  The score varies from 0 to 100 with higher score means severe IBS.
Qualitative difference in patient-reported clinical outcome of Sleep Apnea (Berlin questionnaire) between the 4 groups of subjects included. | At baseline
  It is composed of 3 categories of questions, if 2 or more categories are positive it means a high risk of apnea.
Quantitative difference in Visual Analog Scale (VAS) score for patient's pain between the 4 groups of subjects included. | At baseline
  The score varies from 0 to 100 with higher score means worst pain possible.
Quantitative difference in Visual Analog Scale (VAS) score for patient's fatigue between the 4 groups of subjects included. | At baseline
  The score varies from 0 to 100 with higher score means extreme fatigue.
Quantitative difference in Visual Analog Scale (VAS) score for patient's disease activity between the 4 groups of subjects included. | At baseline
  The score varies from 0 to 100 with higher score means complete Limitation (Unable to Perform Any Activity).
Quantitative difference in Visual Analog Scale (VAS) score for disease activity on the opinion of the physician between the 4 groups of subjects included. | At baseline
  The score varies from 0 to 100 with higher score means complete Limitation (Unable to Perform Any Activity).
Quantitative difference in Pichot Fatigue Scale score between the 4 groups of subjects included. | At baseline
  The score varies from 0 to 32 with higher score means severe fatigue.
Quantitative difference in State-Trait Anxiety Inventory (STAI) score between the 4 groups of subjects included. | At baseline
  The score varies from 20 to 80 with higher score means high anxiety.
Quantitative difference in patient-reported outcome Posttraumatic Stress Disorder Checklist (PCL-5) score between the 4 groups of subjects included, | At baseline
  The score varies from 0 to 80 with higher score means very severe symptoms (Likely posttraumatic stress disorder (PTSD)).
Quantitative difference in patient-reported outcome heath survey Short Form-12 (SF-12) version 2 with Physical Component Summary (PCS) and Mental Component Summary (MCS) scores between the 4 groups of subjects included | At baseline
  The mean is 50 for each score with a standard deviation of 10, a higher score means better health status.
Quantitative difference in Insomnia Severity Index (ISI) score between the 4 groups of subjects included | At baseline
  The score varies from 0 to 28 with higher score means Severe insomnia.
Quantitative difference in Pain Catastrophizing Scale (PCS) score between the 4 groups of subjects included | At baseline
  The score varies from 0 to 52 with higher score means High pain catastrophizing.
Quantitative difference in Rheumatoid factor (FR) auto-antibody level between the 4 groups of subjects included. | At baseline
  Expressed in IU/ml (International Units per Milliliter)
Quantitative difference Anti-Citrullinated Peptide Antibodies (ACPA) level between the 4 groups of subjects included. | At baseline
  Expressed in IU/ml (International Units per Milliliter).
Quantitative difference in C-reactive protein (CRP) level between the 4 groups of subjects included. | At baseline
  Expressed in mg/L (milligram per liter)
Quantitative difference in Neutrophils values between the 4 groups of subjects included. | At baseline
  Expressed in cells/µL (microliter)
Quantitative difference in lymphocytes values between the 4 groups of subjects included. | At baseline
  Expressed in cells/µL (microliter)
Quantitative difference in Platelets (PLT) between the 4 groups of subjects included. | At baseline
  Expressed in platelets/µL (microliter)
Clinical arthritis and Clinically Suspected Arthralgias (CSA). | Baseline, week 26; week 52 and week 104 visit
  Assess the incidence of clinical arthritis in high-risk RA patients overall (group 1 and 2) and in subgroups according to the presence or absence of CSA and the auto-antibody profile at inclusion. The clinical arthritis is detected by the presence of joints swelling in at least 1 of the 44 joints swelling and confirmed by ultrasound.
Quantitative difference in Visual Analog Scale (VAS) score for patient's pain between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline, week 26; week 52 and week 104 visit
  The score varies from 0 to 100 with higher score means worst pain possible. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in Visual Analog Scale (VAS) score for patient's fatigue between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline, week 26; week 52 and week 104 visit
  The score varies from 0 to 100 with higher score means extreme fatigue. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in Visual Analog Scale (VAS) score for patient's disease activity between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline, week 26; week 52 and week 104 visit
  The score varies from 0 to 100 with higher score means complete Limitation (Unable to Perform Any Activity). Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in Visual Analog Scale (VAS) score for disease activity on the opinion of the physician between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline, week 26; week 52 and week 104 visit
  The score varies from 0 to 100 with higher score means complete Limitation (Unable to Perform Any Activity). Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in Pichot Fatigue Scale score between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline, week 26; week 52 and week 104 visit
  The score varies from 0 to 32 with higher score means severe fatigue. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in State-Trait Anxiety Inventory (STAI) score between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline, week 26; week 52 and week 104 visit
  The score varies from 20 to 80 with higher score means high anxiety. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in patient-reported outcome Posttraumatic Stress Disorder Checklist (PCL-5) score between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline, week 26; week 52 and week 104 visit
  The score varies from 0 to 80 with higher score means very severe symptoms (Likely posttraumatic stress disorder (PTSD). Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in patient-reported outcome heath survey Short Form-12 (SF-12) version 2 with Physical Component Summary (PCS) and Mental Component Summary (MCS) scores between the patients who developed clinical arthritis during the 2-year f | Baseline, week 26; week 52 and week 104 visit
  The mean is 50 for each score and a standard deviation of 10, a higher score means better health status. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in Insomnia Severity Index (ISI) score between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline, week 26; week 52 and week 104 visit
  The score varies from 0 to 28 with higher score means Severe insomnia. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in Pain Catastrophizing Scale (PCS) score between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline, week 26; week 52 and week 104 visit
  The score varies from 0 to 52 with higher score means High pain catastrophizing. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in tender joints count between the patients who developed clinical arthritis during the 2-year follow-up and those who did not, among 44 joints across the body. | Baseline, week 26, week 52 and week 104 visit
  The score varies from 0 to 44 with higher score means more active inflammatory joint disease. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in tenosynovitis count between the patients who developed clinical arthritis during the 2-year follow-up and those who did not, among 16 flexor and extensor finger's tendons. | Baseline, week 26, week 52 and week 104 visit
  The score varies from 0 to 44 with higher score means more active inflammatory joint disease. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in difficulties of making a fist between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. Relate this outcome to the risk of developing clinical arthritis. | Baseline, week 26, week 52 and week 104 visit
Quantitative difference in tenosynovitis between the patients who developed clinical arthritis during the 2-year follow-up and those who did not detected by ultrasound. Relate this outcome to the risk of developing clinical arthritis | Baseline, week 26; week 52 and week 104 visit
Quantitative difference in Rheumatoid factor (FR) auto-antibody level between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline, week 26, week 52 and week 104 visit
  Expressed in IU/ml (International Units per Milliliter).Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in Anti-Citrullinated Peptide Antibodies (ACPA) level between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline, week 26, week 52 and week 104 visit
  Expressed in IU/ml (International Units per Milliliter) Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in C-reactive protein (CRP) level between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline, week 26, week 52 and week 104 visit
  Expressed in mg/L (milligram per liter) Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in Neutrophils values between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline, week 26, week 52 and week 104 visit
  Expressed in cells/µL (microliter).Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in lymphocytes values between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline, week 26, week 52 and week 104 visit
  Expressed in cells/µL (microliter). Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in Platelets (PLT) between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline, week 26, week 52 and week 104 visit
  Expressed in platelets/µL (microliter), Relate this outcome to the risk of developing clinical arthritis.
Proportion of patients with ultrasound synovitis in the 2 groups at high-risk of rheumatoid factor (RA) (group 1 and 2). | Baseline, week 26, week 52 and week 104 visit
  Detected by ultrasound in mode B and Doppler on the hand's and feet's articulations with semi-quantitative gradation according to Outcome Measures in Rheumatology (OMERACT) recommendations, between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. Relate this outcome to the risk of developing clinical arthritis.
Proportion of patients with ultrasound tenosynovitis in the 2 groups at high-risk of rheumatoid factor (RA) (group 1 and 2). | Baseline, week 26, week 52 and week 104 visit
  Detected by ultrasound in mode B and Doppler on the hand's and feet's articulations with semi-quantitative gradation according to Outcome Measures in Rheumatology (OMERACT) recommendations, between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. Relate this outcome to the risk of developing clinical arthritis.
Proportion of patients with ultrasound synovitis in the 4 groups of subjects included. | Baseline
  Detected by ultrasound in mode B and Doppler on the hand's and feet's articulations with semi-quantitative gradation according to Outcome Measures in Rheumatology (OMERACT) recommendations. Relate this outcome to the risk of developing clinical arthritis.
Proportion of patients with ultrasound tenosynovitis in the 4 groups of subjects included. | Baseline
  Detected by ultrasound in mode B and Doppler on the hand's and feet's articulations with semi-quantitative gradation according to Outcome Measures in Rheumatology (OMERACT) recommendations. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in synovitis between the 4 groups of subjects included. | Baseline
  Detected by Magnetic Resonance Imaging (MRI) on the dominant hand or the most painful hand. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in bone oedemes between the 4 groups of subjects included. | Baseline
  Detected by Magnetic Resonance Imaging (MRI) on the dominant hand or the most painful hand. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in pinch between the 4 groups of subjects included. | Baseline
  Detected by Magnetic Resonance Imaging (MRI) on the dominant hand or the most painful hand. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in erosion between the 4 groups of subjects included. | Baseline
  Detected by Magnetic Resonance Imaging (MRI) on the dominant hand or the most painful hand. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in tenosynovitis between the 4 groups of subjects included, between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline
  Detected by Magnetic Resonance Imaging (MRI) on the dominant hand or the most painful hand. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in synovitis between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline
  Detected by Magnetic Resonance Imaging (MRI) on the dominant hand or the most painful hand. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in bone oedemes between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline
  Detected by Magnetic Resonance Imaging (MRI) on the dominant hand or the most painful hand. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in pinch between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline
  Detected by Magnetic Resonance Imaging (MRI) on the dominant hand or the most painful hand. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in erosion between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline
  Detected by Magnetic Resonance Imaging (MRI) on the dominant hand or the most painful hand. Relate this outcome to the risk of developing clinical arthritis.
Quantitative difference in tenosynovitis between the patients who developed clinical arthritis during the 2-year follow-up and those who did not. | Baseline
  Detected by Magnetic Resonance Imaging (MRI) on the dominant hand or the most painful hand. Relate this outcome to the risk of developing clinical arthritis.
Analyzing heart rate variability as a risk factor for developing RA | Baseline
  Measurement of heart rate variability in high-risk patients (group 1 + group 2) for RA
Analyze environmental factors associated with the risk of developing clinical arthritis. | Baseline, week 26, week 52 and week 104 visit
  Exposure will be assessed using partial addresses

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: No